CLINICAL TRIAL: NCT06935006
Title: Sonographic Guided Erector Spinae Plane Block Versus Conventional Analgesia After Percutaneous Nephrolithotomy a Comparative Randomized Study
Brief Title: Erector Spinae Block vs Conventional Analgesia for Postoperative Analgesia in PCNL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Azmy, Assistant lecturer of Anaethesia and intensive care unit, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-22-06-35
Record Dates: First submitted 2025-03-09; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Percutaneous Nephrolithotomy (PCNL)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Active Comparator)
  Interventions: Procedure: Sonographic guided Erector spinae plane block
- Conventional analgesia group (Active Comparator)
  Interventions: Drug: Intravenous opioid

INTERVENTIONS:
Procedure: Sonographic guided Erector spinae plane block — Ultrasound guided plane block using 20 ml of 0.25% bupivacaine at the level of transverse process of T8
  Arms: Erector spinae plane block group
Drug: Intravenous opioid — 0.1 mg/kg morphine intravenous pre operative
  Arms: Conventional analgesia group

SUMMARY:
50 adult patients scheduled for percutaneous nephrolithotomy in Sohag university hospitals will be devided in two groups one of them will receive Sonographic guided erector spinae plane block using 20 ml volume of bupivacaine 0.25 percent and the other will receive conventional analgesia of 0.1 mg/kg IV morphine

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to ASA 2 18 to 60 years

Exclusion Criteria:

* patient refusal Significant neurological , psychiatric or neuromascular disease Drug abuse Pregnant or lactating women Suspected coagulopathy Morbid obesity Known allergy to some medications Septicaemia and local infection at block site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of postoperative pain | 1 year
  VAS score for pain measurement